CLINICAL TRIAL: NCT04243083
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single and Multiple Ascending Dose (SAD/MAD) Study in Healthy Subjects To Evaluate The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Of TLL018 Following Oral Administration And With An Open Label Food Effect Panel
Brief Title: A Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Study of TLL018, With Food Effect, in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TLL Pharmaceutical, LLC (Industry)
Responsible Party: Sponsor
Organization: Hangzhou Highlightll Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TLL018-101
Record Dates: First submitted 2020-01-18; First posted 2020-01-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (SAD) (Experimental): There are multiple dose levels or cohorts. Each cohort has 6 subjects randomized to active drugs and 2 subjects randomized to placebo.
  Interventions: Drug: TLL018 tablet, placebo
- Multiple Ascending Dose (MAD) (Experimental): There are multiple dose levels or cohorts. Each cohort has 6 subjects randomized to active drugs and 2 subjects randomized to placebo.
  Interventions: Drug: TLL018 tablet, placebo
- Food Effect Panel (Experimental): Twelve subjects will receive a single dose of TLL018 in 2 treatment periods, one after a high fat, high calorie breakfast (fed) and the second treatment period under fasted conditions to determine the effect of food on the PK of TLL018.
  Interventions: Drug: TLL018 tablet, placebo

INTERVENTIONS:
Drug: TLL018 tablet, placebo — Oral QD

SUMMARY:
TLL018 is developed for treatment of autoimmune and inflammatory diseases including rheumatoid arthritis. The purposes of this study are (1) determining if and at what doses TLL018 is safe and can be tolerated when administered to humans, (2) assessing what TLL018 does to the body and how the body responds to TLL018 when given as single and multiple doses, and (3) assessing potential food effect on TLL018.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are between the ages of 18 and 55 years, inclusive;
3. Female subjects have a negative serum hCG or urine pregnancy test result at screening and Day -1, and meet one of the following criteria:

   1. Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Surgically sterile, with documentation, for at least 3 months prior to screening by one of the following means:

      * Bilateral tubal ligation
      * Bilateral salpingectomy (with or without oophorectomy)
      * Surgical hysterectomy
      * Bilateral oophorectomy (with or without hysterectomy)
   3. Postmenopausal, defined as the following:

      * Last menstrual period greater than 12 months prior to screening
      * Postmenopausal status confirmed by serum follicle stimulating hormone (FSH) and estradiol levels at screening;
4. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs;
5. Normal renal function as determined by Investigator following review of clinical laboratory test results;
6. Non-smoker or no more than 2 tobacco-containing including nicotine replacement products in last 6 months;
7. Body mass index (BMI) of 18.0 to 30.0 kg/m2 inclusive and body weight not less than 50 kg; Subjects with BMI between 30 and 32 kg/m2 may be allowed to participate with the sponsor's approval;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center;
9. Male subjects with female partners of child-bearing potential must agree to use condoms for the duration of the study and until 12 weeks after dosing with the study drug and must refrain from donating sperm for this same period;
10. Ability to swallow and retain oral medication.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Pregnant (as determined by pregnancy test result) and breastfeeding women;
3. Current and/or recent history (<30 days prior to screening and/or <45 days prior to randomization) of a clinically significant bacterial, fungal, parasitic, or mycobacterial infection;
4. Current clinically significant viral infection;
5. Evidence of latent or active tuberculosis, as well as recent exposure or live vaccinations
6. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin;
7. History of pancreatitis or gall stones;
8. History of unexplained syncope, symptomatic hypotension or hypoglycemia;
9. Family history of long QTc syndrome; History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant. QTcF interval >440 msec for males and >460 msec for females;
10. Resting pulse <45 bpm or >100 bpm at screening, only with Day -1 as PI judgement;
11. History of unstable ischemic heart disease or uncontrolled hypertension (blood pressure >140/90 mm Hg at screening, only with Day -1 as PI judgement);
12. History of stomach or intestinal surgery, except that appendectomy and/or cholecystectomy will be allowed;
13. History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance;
14. Poor venous access;
15. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
16. Donated or lost >500 ml of blood in the previous 3 months;
17. Taken any prescription medications within 7 days or 5 half-lives (whichever is longer) of the first dose of study drug;
18. Hospital admission or major surgery within 6 months prior to screening;
19. A history of prescription drug abuse, or illicit drug use within 9 months prior to screening;
20. A history of alcohol abuse according to medical history within 9 months prior to screening;
21. A positive screen for alcohol or drugs of abuse at screening or Day -1;
22. An unwillingness or inability to comply with food and beverage restrictions during study participation;
23. Use of over-the-counter (OTC) medication within 7 days, and herbal (including St John's Wort, herbal teas, garlic extracts) within 7 days prior to dosing (Note: Use of acetaminophen at <2 g/day is permitted until 24 hours prior to dosing);
24. Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study medication with another investigational medication or current enrollment in another investigational drug protocol;
25. Hemoglobin, WBC, or platelet count below the lower reference limit of the testing laboratory. Absolute neutrophil count <2000 cells/uL;
26. Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Number of participants with treatment-emergent adverse events (AEs), serious adverse events (SAEs) and discontinuation due to AEs/SAEs | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Number of adverse events (AEs) according to severity | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Change of blood pressure from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Change of pulse rate from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Change of respiratory rate from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Change of oral temperature from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Number of participants with clinical laboratory abnormalities compared to baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Cohorts: Number of participants with changes in physical examination findings from baseline | Screening up to Day 8 for SAD; Screening up to Day 14 for MAD
Single Ascending Dose (SAD) Cohort: Maximum observed plasma concentration (Cmax) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Time to reach maximum observed plasma concentration (Tmax) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Plasma decay half-life (t1/2) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Area under the curve from time zero to last quantifiable concentration (AUClast) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Mean residence time (MRT) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Apparent clearance (CL/F) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Apparent volume of distribution (Vz/F) of TLL018 | 0 hour (pre-dose - within 60 minutes prior to dosing), and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Maximum observed plasma concentration (Cmax) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Time to reach maximum observed plasma concentration (Tmax) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Plasma decay half-life (t1/2) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Area under the curve from time zero to last quantifiable concentration (AUClast) of TLL018 following oral single ascending dose administration of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Mean residence time (MRT) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Apparent clearance (CL/F) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Apparent volume of distribution (Vz/F) of TLL018 | Day 1 (first dose) at pre-dose, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose; on Days 3 to 6, pre-dose; on Day 7 (last dose): pre-dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Amount of TLL018 recovered unchanged in the urine over the time interval Tau (Aetau) | Day 1 at pre-dose up to 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Percentage of dose of TLL018 recovered unchanged in the urine over the time interval Tau (Aetau %) | Day 1 at pre-dose up to 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Renal clearance (CLr) of TLL018 | Day 1 at pre-dose up to 72 hours post-dose
Food Effect Cohort: Maximum observed plasma concentration (Cmax) of a single oral dose of TLL018 | 0-hour pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Food Effect Cohort: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of a single oral dose of TLL018 | 0-hour pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Food Effect Cohort: Area under the curve from time zero to last quantifiable concentration (AUClast) of a single oral dose of TLL018 | 0-hour pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Food Effect Cohort: Time to reach maximum observed plasma concentration (Tmax) of a single oral dose of TLL018 | 0-hour pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose
Food Effect Cohort: Plasma decay half-life (t1/2) of a single oral dose of TLL018 | 0-hour pre-dose (within 60 minutes prior to dosing) and at 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose

SECONDARY OUTCOMES:
Single Ascending Dose (SAD) Cohort: Changes of white blood cell, neutrophil and lymphocyte counts and platelets from baseline | 0 hour (pre-dose), 4, 8, 12, 24, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Changes of high sensitivity C-reactive protein (hsCRP) and interferon gamma-induced protein 10 (IP-10) concentrations in blood from baseline | 0 hour (pre-dose), 4, 8, 12, 24, 48, and 72 hours post-dose
Single Ascending Dose (SAD) Cohort: Effect on phospho-STAT3 levels in blood cells compared to untreated baseline | 0 hour (pre-dose), 1, 4, 6, 12, 24, and 48 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Changes of white blood cell, neutrophil and lymphocyte counts and platelets from baseline | Day 1 pre-dose, 4, 8, 12 hours post-dose, 24 hours pre-dose, Day 7 pre-dose, 4, 8, 12, 24, 48 and 72 hours post-dose
Multiple Ascending Dose (MAD) Cohort: Changes of high sensitivity C-reactive protein (hsCRP) and interferon gamma-induced protein 10 (IP-10) concentrations in blood from baseline | Day 1 pre-dose, 4, 8, 12 hours post-dose, 24 hours pre-dose, Day 7 pre-dose, 4, 8, 12, 24, 48 and 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Study Director — Frontage Clinical Services
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States